CLINICAL TRIAL: NCT05311735
Title: Autogenous Mineralized and Partial Demineralized Dentin Graft Compared to Freeze Dried Bone Allograft: A Randomized Control Trial
Brief Title: Mineralized and Partial Demineralized Dentin Graft Compared to FDBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Delta Dental Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13712
Record Dates: First submitted 2022-02-21; First posted 2022-04-05 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: * Test group I (mineralized tooth graft): extracted teeth will undergo the mineralization process according to the manufacture's guidelines. Procedure will be done in a specialized equipment for tooth graft preparation (Smart Dentin Grinder® (SDG) (KometaBio), and then sites will be grafted. Remaining graft will be stored appropriately for future grafting in the same patient (according to the guidelines)
  * Test group II (partial-demineralized tooth graft): extracted teeth will be undergone to partial-demineralized process, according to the manufacture's guidelines. Procedures will be done in a specialized equipment for tooth graft preparation (Smart Dentin Grinder® (SDG) (KometaBio), and then sites will be grafted. Remaining graft will be stored appropriately for future grafting in the same patient (according to the guidelines).
  * Control group (FDBA): extracted teeth will be discarded and sites will be grafted with FDBA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Freeze-Dried Bone Allograft Control (Other): -Control group (FDBA): extracted teeth will be discarded and sites will be grafted with FDBA.
  Interventions: Procedure: Freeze-Dried Bone Allograft control
- Mineralized Dentin Graft (Experimental): -Test group I (mineralized tooth graft): extracted teeth will undergo the mineralization process according to the manufacture's guidelines. Procedure will be done in a specialized equipment for tooth graft preparation (Smart Dentin Grinder® (SDG) (KometaBio), and then sites will be grafted. Remaining graft will be stored appropriately for future grafting in the same patient (according to the guidelines)
  Interventions: Procedure: Mineralized Dentin Graft
- Partial-Demineralized Dentin Graft (Experimental): -Test group II (partial-demineralized tooth graft): extracted teeth will be undergone to partial-demineralized process, according to the manufacture's guidelines. Procedures will be done in a specialized equipment for tooth graft preparation (Smart Dentin Grinder® (SDG) (KometaBio), and then sites will be grafted. Remaining graft will be stored appropriately for future grafting in the same patient (according to the guidelines).
  Interventions: Procedure: Partial-Demineralized Dentin Graft

INTERVENTIONS:
Procedure: Freeze-Dried Bone Allograft control — Bone grafting to prevent alveolar ridge collapse after tooth removal
  Arms: Freeze-Dried Bone Allograft Control
Procedure: Mineralized Dentin Graft — Mineralized tooth graft used as a bone graft substitute to prevent alveolar ridge collapse after tooth removal
  Arms: Mineralized Dentin Graft
Procedure: Partial-Demineralized Dentin Graft — Partially mineralized tooth graft used as a bone graft substitute to prevent alveolar ridge collapse after tooth removal
  Arms: Partial-Demineralized Dentin Graft

SUMMARY:
The bone grafting materials currently used in dentistry are autografts, allografts, xenografts, and alloplastic grafts. Among these different types of bone graft materials, autografts are considered to have the most predictable results due to its properties of osteogenesis, osteoinduction and osteoconduction. However, bone autografts are rarely used due to the high morbidity associated with harvesting the bone graft from the patient with a second surgical site. Because of the increased risk to the patient with autogenous bone grafts, the current standard of care is an allograft, which is a bone graft harvested from cadaver sources such as Freeze-Dried Bone Allograft (FDBA). While allografts can only possess the qualities of osteoinduction and osteoconduction, they also have dramatically less morbidity due to the lack of a second surgical site.

Studies have shown that autogenous dentin grafts promote all three ideal mechanisms for bone regeneration. There are two methods to generate autogenous dentin grafts. One is to collect the extracted tooth and to send it to a tooth bank for the preparation process. The second is to process the extracted tooth in a clinical setting chairside, for a graft. A dentin graft can undergo different treatments such as demineralization, mineralization, and partial-demineralization. Although the autogenous dentin graft has shown positive results for bone regeneration, the comparison between partial-demineralized, mineralized autogenous dentin grafts, and freeze-dried bone grafts in the clinical setting for immediate grafting has not been studied in humans. Thus, there is a need to study the benefits of autogenous dentin partial-demineralized and mineralized grafts versus freeze-dried bone allografts regarding clinical, radiographically (bone volume and density), and efficacy results. This research addresses these areas of need.

DETAILED DESCRIPTION:
The bone grafting materials currently used in dentistry are autografts, allografts, xenografts, and alloplastic grafts. Among these different types of bone graft materials, autografts are considered to have the most predictable results due to its properties of osteogenesis, osteoinduction and osteoconduction. However, bone autografts are rarely used due to the high morbidity associated with harvesting the bone graft from the patient with a second surgical site. Because of the increased risk to the patient with autogenous bone grafts, the current standard of care is an allograft, which is a bone graft harvested from cadaver sources such as Freeze-Dried Bone Allograft (FDBA). While allografts can only possess the qualities of osteoinduction and osteoconduction, they also have dramatically less morbidity due to the lack of a second surgical site.

Studies have shown that autogenous dentin grafts promote all three ideal mechanisms for bone regeneration. There are two methods to generate autogenous dentin grafts. One is to collect the extracted tooth and to send it to a tooth bank for the preparation process. The second is to process the extracted tooth in a clinical setting chairside, for a graft. A dentin graft can undergo different treatments such as demineralization, mineralization, and partial-demineralization. Although the autogenous dentin graft has shown positive results for bone regeneration, the comparison between partial-demineralized, mineralized autogenous dentin grafts, and freeze-dried bone grafts in the clinical setting for immediate grafting has not been studied in humans. Thus, there is a need to study the benefits of autogenous dentin partial-demineralized and mineralized grafts versus freeze-dried bone allografts regarding clinical, radiographically (bone volume and density), and efficacy results. This research addresses these areas of need.

A. Specific Aims

Specific Aim 1:

Is there a clinical-radiographical difference in terms of bone volume and density between mineralized dentin grafts, partial demineralized tooth grafts, and FDBA?

Null Hypothesis (Ho): Experimental groups (Mineralized, and partial demineralized dentin grafts) do not have positive changes in terms of bone volume and density when compared to FDBA

Alternative Hypothesis (H1): Experimental groups (Mineralized, and partial demineralized dentin grafts) show better results in terms of bone volume and density when compared to FDBA.

Secondary Aim:

Evaluate if there is any difference in terms of efficacy among partial-demineralized dentin graft, mineralized dentin graft and FDBA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old
* Able to understand and sign a written informed consent form and willing to fulfil all study requirements.
* Alveolar sockets with intact four-wall architecture.
* Patients with at least a tooth that need to be extracted.

Exclusion Criteria:

* Uncontrolled systemic disease
* Currently smoking >10 cigarettes per day
* History of head and/or neck radiotherapy in the past five years
* Bisphosphonates current use or history of IV bisphosphonate
* Pregnant, expecting to become pregnant, or lactating women.
* Presence of active periodontal disease.
* Teeth that underwent root canal fillings
* Teeth with acute infection at the site of extraction.
* Teeth with periapical infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Clinical-radiographical differences in terms of bone volume between dentin tooth grafts and FDBA. | 6 months post guided bone regeneration procedure
  Is there a clinical-radiographical difference in terms of bone volume between mineralized dentin grafts, partial demineralized tooth grafts and FDBA, as measured in millimeters, with calibrated devices?
Clinical-radiographical differences in terms of bone density between dentin tooth grafts and FDBA. | 6 months post guided bone regeneration procedure
  Is there a clinical-radiographical difference in terms of bone density between mineralized dentin grafts, partial demineralized tooth grafts and FDBA, as measured with Hounsfield Units?

SECONDARY OUTCOMES:
Surgical efficiency utilizing dentin tooth graft and FDBA. | 6 months post guided bone regeneration procedure
  Is there any difference in terms of surgical efficiency among partial-demineralized tooth graft, mineralized tooth graft and FDBA, as determined by length of time of surgical procedure?
Surgical cost saving measurement utilizing dentin tooth graft and FDBA. | 6 months post guided bone regeneration procedure
  Is there any difference in terms of surgical cost savings among partial-demineralized tooth graft, mineralized tooth graft and FDBA, as determined by length of time of surgical procedure, as measured by the total overhead expended per procedure type?

CONTACTS AND LOCATIONS:
Overall Officials: Robin Henderson, DMD MS, Principal Investigator — University of Oklahoma College of Dentistry
Locations (1):
- University of Oklahoma College of Dentistry Graduate Periodontics, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
It is estimated that individual patient date will be shared to a very limited number of individuals to help with facilitating the statistical analysis of the study, as well as writing up the Master Thesis and future publications. Also, upon request, it is required to share study related information to our internal Institutional Review Board.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The estimated time frame for sharing data would be approximately until May 2025
Access Criteria: Institutional Review Board officials, Master Thesis Chair and Committee members, and statisticians, will be able to review data. Also, Dr. John Corbett, will be performing a followup study and possibly extending the time frame for Dr. Perozo's study measurement. It is also anticipated, but not actual, that future studies be performed for longitudinal analysis.

REFERENCES:
- [Background] Jung RE, Fenner N, Hammerle CH, Zitzmann NU. Long-term outcome of implants placed with guided bone regeneration (GBR) using resorbable and non-resorbable membranes after 12-14 years. Clin Oral Implants Res. 2013 Oct;24(10):1065-73. doi: 10.1111/j.1600-0501.2012.02522.x. Epub 2012 Jun 15. PMID 22697628
- [Background] Ike M, Urist MR. Recycled dentin root matrix for a carrier of recombinant human bone morphogenetic protein. J Oral Implantol. 1998;24(3):124-32. doi: 10.1563/1548-1336(1998)0242.3.CO;2. PMID 9893518
- [Background] Saygin NE, Tokiyasu Y, Giannobile WV, Somerman MJ. Growth factors regulate expression of mineral associated genes in cementoblasts. J Periodontol. 2000 Oct;71(10):1591-600. doi: 10.1902/jop.2000.71.10.1591. PMID 11063392
- [Background] Emecen P, Akman AC, Hakki SS, Hakki EE, Demiralp B, Tozum TF, Nohutcu RM. ABM/P-15 modulates proliferation and mRNA synthesis of growth factors of periodontal ligament cells. Acta Odontol Scand. 2009;67(2):65-73. doi: 10.1080/00016350802555525. PMID 19031159
- [Background] Kim YK, Kim SG, Byeon JH, Lee HJ, Um IU, Lim SC, Kim SY. Development of a novel bone grafting material using autogenous teeth. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Apr;109(4):496-503. doi: 10.1016/j.tripleo.2009.10.017. Epub 2010 Jan 8. PMID 20060336
- [Background] Kim YK, Kim SG, Yun PY, Yeo IS, Jin SC, Oh JS, Kim HJ, Yu SK, Lee SY, Kim JS, Um IW, Jeong MA, Kim GW. Autogenous teeth used for bone grafting: a comparison with traditional grafting materials. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Jan;117(1):e39-45. doi: 10.1016/j.oooo.2012.04.018. Epub 2012 Aug 30. PMID 22939321
- [Background] Koga T, Minamizato T, Kawai Y, Miura K, I T, Nakatani Y, Sumita Y, Asahina I. Bone Regeneration Using Dentin Matrix Depends on the Degree of Demineralization and Particle Size. PLoS One. 2016 Jan 21;11(1):e0147235. doi: 10.1371/journal.pone.0147235. eCollection 2016. PMID 26795024
- [Background] Binderman, Itzhak, Gideon Hallel, Casap Nardy, Avinoam Yaffe, and Lari Sapoznikov.
- [Background] Phillips DJ, Swenson DT, Johnson TM. Buccal bone thickness adjacent to virtual dental implants following guided bone regeneration. J Periodontol. 2019 Jun;90(6):595-607. doi: 10.1002/JPER.18-0304. Epub 2019 Jan 10. PMID 30578550